CLINICAL TRIAL: NCT04055961
Title: Atrial Fibrillation Ablation Registry Protocol Number: 3122-2016
Brief Title: Atrial Fibrillation Ablation Registry
Acronym: AFib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Colleen Balius, Clinical Data Coordinator, Hoag Memorial Hospital Presbyterian
Other Study IDs: 171-19-CV
Record Dates: First submitted 2019-08-08; First posted 2019-08-14 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Atrial Fibrillation Ablation — A procedure used to treat an irregular heart rhythm (arrhythmia)

SUMMARY:
The Atrial Fibrillation Ablation Registry (AFib Ablation Registry™) is designed to assess the prevalence, demographics, management, and outcomes of patients undergoing percutaneous catheter ablation procedures to treat atrial fibrillation (AF).

DETAILED DESCRIPTION:
The Atrial Fibrillation Ablation Registry (AFib Ablation Registry™) is designed to assess the prevalence, demographics, management, and outcomes of patients undergoing percutaneous catheter ablation procedures to treat atrial fibrillation (AF). Patient-level data will be submitted by participating hospitals on a quarterly basis to the American College of Cardiology Foundation's National Cardiovascular Data Registry (NCDR™). The primary aims of the AFib Ablation Registry are to optimize the outcomes and management of patients through the implementation of evidence-based guideline recommendations in clinical practice, facilitate efforts to improve the quality and safety for patients undergoing percutaneous catheter ablation procedures, investigate novel quality improvement methods and provide risk-adjusted assessment of patients for comparison with nationwide NCDR data. The secondary purpose of the AFib Ablation Registry is to serve as a rich source of clinical data to support assessments of short- and long-term safety, comparative and cost effectiveness research, and as a scalable data infrastructure for post market studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. 18 years and older
3. Undergoing percutaneous catheter ablation procedures to treat atrial fibrillation

Exclusion Criteria:

1. none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, 18 years and older, undergoing percutaneous catheter ablation procedures to treat atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Unsuccessful treatment rate | 1 year
  measured by the number of repeated procedure

SECONDARY OUTCOMES:
Adverse Events | 1 year
  Number of participants with adverse events that are related to treatment (i.e. cardiac tamponade, periprocedural stroke, pulmonary vein stenosis, esophageal damage, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Leila Andres, Study Chair — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoah Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No